CLINICAL TRIAL: NCT04212559
Title: Hemodynamic Effects of Negative Pressure Ventilation in Chronic Obstructive Pulmonary Disease Assessed Using Non-Invasive Electrical Cardiometry
Brief Title: Hemodynamic Effects of Negative Pressure Ventilation in Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: Fu Jen Catholic University (Other)
Responsible Party: Principal Investigator, Ke-Yun, Chao, Head of Respiratory Therapist, Fu Jen Catholic University
Other Study IDs: C107137
Record Dates: First submitted 2019-11-16; First posted 2019-12-27 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2019-11

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NPV group: Patients who had treated in pulmonary rehabilitation unit with NPV
  Interventions: Other: Received negative pressure ventilation

INTERVENTIONS:
Other: Received negative pressure ventilation — Patients who received a negative pressure during inspiratory phase.

SUMMARY:
Negative pressure ventilation (NPV) is a non-invasive ventilation mode which provide better lung expansion. The major complication of NPV is decrease blood pressure and affects the hemodynamics. The effects of NPV on chronic obstructive pulmonary disease (COPD) patients with pulmonary rehabilitation program remains unknown.

DETAILED DESCRIPTION:
Both of NPV or positive pressure ventilation (PPV) has impact of hemodynamics. NPV with cuirass ventilator increases venous return and leads to ventricular filling and increases cardiac output (CO); In contrast to NPV, the effect of PPV in most situations is a decreased venous return and leads to decreased CO. NPV improving ventilation and work of breathing in patients with chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* Patients with COPD who received pulmonary rehabilitation program with NPV treatment

Exclusion Criteria:

* Recent exacerbation within 3-months
* Existing of tracheostomy
* Absence of NPV used
* Required of oxygen supplement during NPV
* Diagnosed of neuromuscular disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
CO (cardiac output) | 20 minutes
  Change of Cardiac output before and after NPV treatment
SV (stroke volume) | 20 minutes
  Change of stroke volume before and after NPV treatment

SECONDARY OUTCOMES:
SpO2 | 20 minutes
  Change of oxygen saturation before and after NPV treatment
RR (respiratory rate) | 20 minutes
  Change of respiratory rate before and after NPV treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Fu Jen Catholic University Hospital, Fu Jen Catholic University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No